CLINICAL TRIAL: NCT03472885
Title: A Phase 2 Open-label Study of ACH-0144471 in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Who Have an Inadequate Response to Eculizumab Monotherapy
Brief Title: Study of Danicopan in Participants With Paroxysmal Nocturnal Hemoglobinuria With Inadequate Response to Eculizumab
Acronym: PNH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACH471-101; 2016-003526-16 (EudraCT Number); U1111-1209-4655 (Other: UTN)
Record Dates: First submitted 2018-03-15; First posted 2018-03-21 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: PNH; Paroxysmal Nocturnal Hemoglobinuria; ACH-0144471; Danicopan; Eculizumab; ALXN2040
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — danicopan; eculizumab

STUDY DESIGN:
Intervention Model Description: Four groups will be studied and enrolled sequentially.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: 100 mg Danicopan TID + Eculizumab (Experimental): Starting dose of 100 mg danicopan TID in combination with eculizumab.
  Interventions: Drug: Danicopan; Drug: Eculizumab
- Group 2: Initial dose 100 or 150 mg Danicopan TID + Eculizumab (Experimental): Starting dose of 100 or 150 mg danicopan TID in combination with eculizumab.
  Interventions: Drug: Danicopan; Drug: Eculizumab
- Group 3: Initial dose of 100, 150, or 200 mg Danicopan TID + Eculizumab (Experimental): Starting dose of 100, 150, or 200 mg danicopan TID in combination with eculizumab.
  Interventions: Drug: Danicopan; Drug: Eculizumab
- Group 4: Optimal Dose of Danicopan TID + Eculizumab (Experimental): Optimal dose (starting dose of either 100, 150, or 200 mg, as determined from Groups 1-3) of danicopan TID in combination with eculizumab.
  Interventions: Drug: Danicopan; Drug: Eculizumab

INTERVENTIONS:
Drug: Danicopan — Participants received a daily oral dose of danicopan TID during the treatment period.
Drug: Eculizumab — Participants received intravenous eculizumab administered at the participant's usual dose and schedule.
  Other Names: Soliris

SUMMARY:
To determine the effectiveness of ACH-0144471 (also known as danicopan and ALXN2040) in improving anemia when given with eculizumab for 24 weeks in participants with PNH. Danicopan dose may be increased within each participant, to a maximum of 200 milligrams (mg) three times daily (TID) based on safety and efficacy at protocol-specified time points.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness of danicopan in improving anemia, as measured by increased blood hemoglobin, when given with eculizumab (a drug commonly used for treatment of PNH) for 24 weeks in participants with PNH.

The 24-week treatment period was followed by a long-term extension phase. In the extension phase, participants received the same danicopan dose plus eculizumab as they were receiving at the end of 24-week treatment phase.

Results are reported for the 24-week treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with PNH
* Have received at least one red blood cell transfusion within last 12 weeks
* Anemia with adequate reticulocytosis
* Must be on a stable regimen of eculizumab
* Platelet count ≥ 40,000/microliter without the need for platelet transfusions
* Documentation of vaccination for Neisseria meningitidis, Haemophilus influenza, and Streptococcus pneumoniae or willingness to receive vaccinations based on local guidelines
* Willingness to receive antibiotic prophylaxis
* Female participants must use highly effective birth control to prevent pregnancy during the clinical trial and for 30 days after their last dose of study drug
* Male participants must use a highly effective birth control with a female partner to prevent pregnancy during the clinical trial and for 90 days after the last dose of study drug

Key Exclusion Criteria:

* Current evidence of bone marrow failure or aplastic anemia requiring treatment
* History of a major organ transplant or hematopoietic stem cell/marrow transplant
* Received another investigational agent within 30 days or 5 half-lives of the investigational agent prior to study entry, whichever is greater
* Documented C5 complement protein mutations
* Known or suspected complement deficiency
* Contraindication to any of the required vaccinations
* Active bacterial infection or clinically significant active viral infection, a body temperature >38°C, or other evidence of infection
* History of meningococcal infection, or a first-degree relative or household contact with a history of meningococcal infection
* History of hypersensitivity reactions to commonly used antibacterial agents

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Clinical Study Site, Baltimore, Maryland
  - Clinical Study Site, Cleveland, Ohio
- Italy (2):
  - Clinical Study Site, Florence
  - Clinical Study Site, Naples
- Clinical Study Site, London, United Kingdom

REFERENCES:
- [Derived] Kulasekararaj AG, Risitano AM, Maciejewski JP, Notaro R, Browett P, Lee JW, Huang M, Geffner M, Brodsky RA. Phase 2 study of danicopan in patients with paroxysmal nocturnal hemoglobinuria with an inadequate response to eculizumab. Blood. 2021 Nov 18;138(20):1928-1938. doi: 10.1182/blood.2021011388. PMID 34314483

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a 24-Week Treatment Period and Long-term Extension (LTE) Period.
Groups:
- Danicopan + Eculizumab: Participants were administered 100, 150, or 200 milligrams (mg) danicopan three times daily (TID) in combination with eculizumab for 24 weeks. Danicopan dose may have been increased within each participant, to a maximum of 200 mg TID based on safety and efficacy. After completing the 24-Week Treatment Period, participants who received clinical benefit (as assessed by the Investigator based on improvement in hemoglobin) continued into the LTE and received the same dose of danicopan plus eculizumab treatment as that received at the end of the 24-Week Treatment Period.
Period: 24-Week Treatment Period
Arm/Group | Danicopan + Eculizumab
Started | 12
Safety Population: Received at Least 1 Dose of Study Drug | 12
Efficacy Population: Received Study Drug for at Least 4 Weeks | 11
Completed | 11
Not Completed | 1
Not completed — Adverse Event | 1
Period: LTE Period (Maximum Exposure: 1463 Days)
Arm/Group | Danicopan + Eculizumab
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: Received at least 1 dose of study drug.
Groups:
- Danicopan + Eculizumab: Participants were administered 100, 150, or 200 mg danicopan TID in combination with eculizumab for 24 weeks. Danicopan dose may have been increased within each participant, to a maximum of 200 mg TID based on safety and efficacy. After completing the 24-Week Treatment Period, participants who received clinical benefit (as assessed by the Investigator based on improvement in hemoglobin) continued into the LTE and received the same dose of danicopan plus eculizumab treatment as that received at the end of the 24-Week Treatment Period.
Arm/Group | Danicopan + Eculizumab
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.59 (16.385)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7
  Asian | 1
  Black or African American | 3
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Hemoglobin At Week 24
Time Frame: Baseline, Week 24
Population: Efficacy Population: All treated participants who received at least 4 weeks of danicopan.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Danicopan + Eculizumab
Number analyzed (Participants) | 11
g/dL
  Baseline | 7.94 (1.425)
  Week 24 | 10.33 (1.661)
  Change from Baseline | 2.39 (1.333)

2. Secondary Outcome: Number Of Units Of Red Blood Cells (RBCs) Transfused During 24 Weeks Of Treatment
Time Frame: Within 24 weeks prior to first dose and during 24-week treatment period
Population: Efficacy Population: All treated participants who received at least 4 weeks of danicopan.
Measure: Mean (Standard Deviation); unit: RBC units
Arm/Group | Danicopan + Eculizumab
Number analyzed (Participants) | 11
RBC units
  Within 24 Weeks Prior to First Dose | 4.5 (3.96)
  During 24-Week Treatment Period | 0.2 (0.60)

3. Secondary Outcome: Number Of Participants Without RBC Transfusions During 24 Weeks Of Treatment
Time Frame: Within 24 weeks prior to first dose and during 24-week treatment period
Population: Efficacy Population: All treated participants who received at least 4 weeks of danicopan.
Measure: Count of Participants; unit: Participants
Arm/Group | Danicopan + Eculizumab
Number analyzed (Participants) | 11
Participants
  Within 24 Weeks Prior to First Dose | 1
  During 24-Week Treatment Period | 10

4. Secondary Outcome: Change From Baseline In Lactate Dehydrogenase At Week 24
Time Frame: Baseline, Week 24
Population: Efficacy Population: All treated participants who received at least 4 weeks of danicopan.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Danicopan + Eculizumab
Number analyzed (Participants) | 11
IU/L
  Baseline | 244.5 (74.40)
  Week 24 | 239.5 (48.48)
  Change from Baseline | -5.0 (48.60)

5. Secondary Outcome: Number Of Participants With Serious Adverse Events (SAEs), Grade 3 And Grade 4 Adverse Events (AEs), And Events Leading To Discontinuation Of Study Drug
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), important medical event or reaction. The intensity of an AE was graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Adverse Event Severity Grading Table. A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 (after dosing) through end of study (maximum exposure: 1631 days)
Population: Participants who received at least 1 dose of danicopan were included in the safety assessment.
Measure: Count of Participants; unit: Participants
Groups:
- 24-Week Treatment Period: Danicopan + Eculizumab: Participants were administered 100, 150, or 200 mg danicopan TID in combination with eculizumab for 24 weeks. Danicopan dose may have been increased within each participant, to a maximum of 200 mg TID based on safety and efficacy.
- LTE Period: Danicopan + Eculizumab: After completing the 24-Week Treatment Period, participants who received clinical benefit (as assessed by the Investigator based on improvement in hemoglobin) continued into the LTE and received the same dose of danicopan plus eculizumab treatment as that received at the end of the 24-Week Treatment Period.
Arm/Group | 24-Week Treatment Period: Danicopan + Eculizumab | LTE Period: Danicopan + Eculizumab
Number analyzed (Participants) | 12 | 11
Participants
  SAEs | 2 | 7
  Grade 3 AEs | 4 | 6
  Grade 4 AEs | 1 | 1
  AEs Leading to Discontinuation of Study Drug | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through end of study (maximum exposure: 1631 days)
Description: Participants who received at least 1 dose of danicopan were included in the safety assessment.
Arm/Group | 24-Week Treatment Period: Danicopan + Eculizumab | LTE Period: Danicopan + Eculizumab
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/12 | 7/11
Other Adverse Events (participants affected / at risk) | 10/12 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 24-Week Treatment Period: Danicopan + Eculizumab (N=12) | LTE Period: Danicopan + Eculizumab (N=11)
Pneumonia (Infections and infestations) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Tracheobronchitis viral (Infections and infestations) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemoglobinuria (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 24-Week Treatment Period: Danicopan + Eculizumab (N=12) | LTE Period: Danicopan + Eculizumab (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Palpitations (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Periorbital swelling (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 2 | 3
Feeling abnormal (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 4
Thirst (General disorders) | 1 | 0
Vaccination site pain (General disorders) | 2 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 5
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Fibrin D dimer increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 5
Anxiety (Psychiatric disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
COVID-19 (Infections and infestations) | 0 | 6
Conjunctivitis (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Pain (General disorders) | 0 | 2
Chest discomfort (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 1
Anosmia (Nervous system disorders) | 0 | 2
Ageusia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gingival discomfort (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Saliva altered (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Transfusion-associated dyspnoea (Injury, poisoning and procedural complications) | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Immunisation reaction (Immune system disorders) | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemoglobinuria (Renal and urinary disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Disturbance in attention (Nervous system disorders) | 1 | 1
Influenza like illness (General disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT03472885/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT03472885/SAP_001.pdf